CLINICAL TRIAL: NCT02892136
Title: Technical Development for Pediatric Cardiovascular MRI
Status: Active, not recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Russell Cross, MD, Children's National Research Institute
Other Study IDs: 2359
Record Dates: First submitted 2016-07-21; First posted 2016-09-08 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Congenital Heart Disease; Cardiovascular Disease
MeSH Terms: conditions — Heart Defects, Congenital; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will explore new ways of using magnetic resonance imaging (MRI) to evaluate pediatric patients with cardiovascular disease,congenital heart disease in patients of all ages, fetuses undergoing clinically indicated MR imaging.

DETAILED DESCRIPTION:
The purpose of this protocol is to allow development and testing of new MRI techniques suitable for evaluating patients with cardiovascular disease, congenital heart disease, fetal cardiac structure, function, and physiology, and other fetal organ analysis. Individuals referred to Children's National Medical Center for a clinically indicated cardiac MRI or cardiac catheterization by their primary referring cardiologist or obstetrician, and who are enrolled in this study may also undergo additional research imaging.

Since such technical development work often depends on preliminary studies in healthy volunteers, the protocol also recruits healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Clinically indicated exams

1. Patients who are undergoing a medically indicated MRI scan or cardiac catheterization procedure
2. Patients who are medically judged to have no contraindications to MRI scan
3. Age inclusion: infant to adult
4. Written informed consent and assent, when applicable

Volunteers

1. Written informed consent from any normal volunteer 8 years of age or older for a noncontrast, nonsedated cardiac MRI
2. Normal adult volunteer to undergo cardiac MRI with contrast agent

Fetal exams

1. Age inclusion:18 years and older
2. Second or third trimester (greater than 13 weeks)

Exclusion Criteria:

1. All patients who are medically judged to have contraindication(s) to MRI scanning will be excluded. Contraindications include implanted metal devices which are contraindicated for MRI scanning:

   * Central nervous system aneurysm clips;
   * Implanted neural stimulator;
   * Implanted cardiac pacemaker or defibrillator;
   * Cochlear implant;
   * Ocular foreign body (e.g. metal shavings);
   * Implanted Insulin pump;
   * Metal shrapnel or bullet.
2. Exclusion criteria for Bicycle Stress MRI

   * Myocardial infarction within 24 hours
   * Active myocarditis
   * Uncontrolled heart failure
   * Severe left ventricular outflow tract obstruction
3. Exclusion Criteria for adult volunteers undergoing MRI with administration of contrast agent:

   * 60 years of age or older
   * Renal Disease; Glomerular Filtration rate (eGFR < 30 ml/min/1.73 m2) will be determined by a simple blood test done at the bedside
   * Use of diuretics
   * Diagnosis of hypertension and diabetes
4. Exclusion criteria for volunteers undergoing both contrast and non-contrast

   MRI scans:
   * Pregnant women:

     1. Women of childbearing potential will be required to have a screening urine pregnancy test
5. Exclusion criteria for

   * Pregnant woman for whom 15 additional minutes lying flat in the MR scanner would represent a risk (i.e. severe claustrophobia, congestive heart failure)
   * Pregnant minor under the age of 18
   * Less than 13 weeks gestation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals referred to Children's National Medical Center for a clinically indicated cardiac MRI or cardiac catheterization by their primary referring cardiologist will be considered potential candidates for inclusion in technical development research.
  Technical development work often depends on preliminary studies in healthy volunteers. This protocol also enrolls healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate innovative noninvasive MRI techniques suitable for evaluating pediatric patients with cardiovascular disease, congenital cardiac disease, and fetal organ analysis including cardiac structure, function, and physiology. | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Natural history of congenital heart disease | through study completion, an average of 1 year
  A secondary objective of this protocol is to catalog results from MR imaging studies that can be used to describe the natural history of congenital heart disease and other cardiovascular diseases acquired in the young.

CONTACTS AND LOCATIONS:
Overall Officials: Russell R Cross, MD, Principal Investigator — Children's National Health Systems
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beerbaum P, Sarikouch S, Laser KT, Greil G, Burchert W, Korperich H. Coronary anomalies assessed by whole-heart isotropic 3D magnetic resonance imaging for cardiac morphology in congenital heart disease. J Magn Reson Imaging. 2009 Feb;29(2):320-7. doi: 10.1002/jmri.21655. PMID 19161183
- [Background] Didier D, Ratib O, Beghetti M, Oberhaensli I, Friedli B. Morphologic and functional evaluation of congenital heart disease by magnetic resonance imaging. J Magn Reson Imaging. 1999 Nov;10(5):639-55. doi: 10.1002/(sici)1522-2586(199911)10:53.0.co;2-l. PMID 10548772
- [Background] Frakes DH, Smith MJ, Parks J, Sharma S, Fogel SM, Yoganathan AP. New techniques for the reconstruction of complex vascular anatomies from MRI images. J Cardiovasc Magn Reson. 2005;7(2):425-32. doi: 10.1081/jcmr-200053637. PMID 15881525
- [Background] Krishnamurthy R. Pediatric cardiac MRI: anatomy and function. Pediatr Radiol. 2008 May;38 Suppl 2:S192-9. doi: 10.1007/s00247-008-0786-0. No abstract available. PMID 18401610
- [Background] Sarikouch S, Peters B, Gutberlet M, Leismann B, Kelter-Kloepping A, Koerperich H, Kuehne T, Beerbaum P. Sex-specific pediatric percentiles for ventricular size and mass as reference values for cardiac MRI: assessment by steady-state free-precession and phase-contrast MRI flow. Circ Cardiovasc Imaging. 2010 Jan;3(1):65-76. doi: 10.1161/CIRCIMAGING.109.859074. Epub 2009 Oct 9. PMID 19820203
- [Background] Uribe S, Muthurangu V, Boubertakh R, Schaeffter T, Razavi R, Hill DL, Hansen MS. Whole-heart cine MRI using real-time respiratory self-gating. Magn Reson Med. 2007 Mar;57(3):606-13. doi: 10.1002/mrm.21156. PMID 17326164
- [Background] Valverde I, Parish V, Tzifa A, Head C, Sarikouch S, Greil G, Schaeffter T, Razavi R, Beerbaum P. Cardiovascular MR dobutamine stress in adult tetralogy of Fallot: disparity between CMR volumetry and flow for cardiovascular function. J Magn Reson Imaging. 2011 Jun;33(6):1341-50. doi: 10.1002/jmri.22573. PMID 21591002
- [Background] Beerbaum P, Korperich H, Barth P, Esdorn H, Gieseke J, Meyer H. Noninvasive quantification of left-to-right shunt in pediatric patients: phase-contrast cine magnetic resonance imaging compared with invasive oximetry. Circulation. 2001 May 22;103(20):2476-82. doi: 10.1161/01.cir.103.20.2476. PMID 11369688
- [Background] Beerbaum P, Korperich H, Gieseke J, Barth P, Peuster M, Meyer H. Rapid left-to-right shunt quantification in children by phase-contrast magnetic resonance imaging combined with sensitivity encoding (SENSE). Circulation. 2003 Sep 16;108(11):1355-61. doi: 10.1161/01.CIR.0000087603.97036.C2. Epub 2003 Aug 25. PMID 12939211
- [Background] Bell A, Beerbaum P, Greil G, Hegde S, Toschke AM, Schaeffter T, Razavi R. Noninvasive assessment of pulmonary artery flow and resistance by cardiac magnetic resonance in congenital heart diseases with unrestricted left-to-right shunt. JACC Cardiovasc Imaging. 2009 Nov;2(11):1285-91. doi: 10.1016/j.jcmg.2009.07.009. PMID 19909932
- [Background] Korperich H, Gieseke J, Barth P, Hoogeveen R, Esdorn H, Peterschroder A, Meyer H, Beerbaum P. Flow volume and shunt quantification in pediatric congenital heart disease by real-time magnetic resonance velocity mapping: a validation study. Circulation. 2004 Apr 27;109(16):1987-93. doi: 10.1161/01.CIR.0000126494.66859.A2. Epub 2004 Apr 5. PMID 15066942
- [Background] Uribe S, Beerbaum P, Sorensen TS, Rasmusson A, Razavi R, Schaeffter T. Four-dimensional (4D) flow of the whole heart and great vessels using real-time respiratory self-gating. Magn Reson Med. 2009 Oct;62(4):984-92. doi: 10.1002/mrm.22090. PMID 19672940
- [Background] Hansen MS, Kozerke S, Pruessmann KP, Boesiger P, Pedersen EM, Tsao J. On the influence of training data quality in k-t BLAST reconstruction. Magn Reson Med. 2004 Nov;52(5):1175-83. doi: 10.1002/mrm.20256. PMID 15508162
- [Background] Lardo AC. Real-time magnetic resonance imaging: diagnostic and interventional applications. Pediatr Cardiol. 2000 Jan-Feb;21(1):80-98. doi: 10.1007/s002469910010. PMID 10672617
- [Background] Muthurangu V, Lurz P, Critchely JD, Deanfield JE, Taylor AM, Hansen MS. Real-time assessment of right and left ventricular volumes and function in patients with congenital heart disease by using high spatiotemporal resolution radial k-t SENSE. Radiology. 2008 Sep;248(3):782-91. doi: 10.1148/radiol.2482071717. Epub 2008 Jul 15. PMID 18632528
- [Background] Parish V, Hussain T, Beerbaum P, Greil G, Nagel E, Razavi R, Schaeffter T, Uribe S. Single breath-hold assessment of ventricular volumes using 32-channel coil technology and an extracellular contrast agent. J Magn Reson Imaging. 2010 Apr;31(4):838-44. doi: 10.1002/jmri.22061. PMID 20373427
- [Background] Sorensen TS, Korperich H, Greil GF, Eichhorn J, Barth P, Meyer H, Pedersen EM, Beerbaum P. Operator-independent isotropic three-dimensional magnetic resonance imaging for morphology in congenital heart disease: a validation study. Circulation. 2004 Jul 13;110(2):163-9. doi: 10.1161/01.CIR.0000134282.35183.AD. Epub 2004 Jun 21. PMID 15210590
- [Background] Su JT, Chung T, Muthupillai R, Pignatelli RH, Kung GC, Diaz LK, Vick GW 3rd, Kovalchin JP. Usefulness of real-time navigator magnetic resonance imaging for evaluating coronary artery origins in pediatric patients. Am J Cardiol. 2005 Mar 1;95(5):679-82. doi: 10.1016/j.amjcard.2004.10.051. PMID 15721121
- [Background] Kul S, Korkmaz HA, Cansu A, Dinc H, Ahmetoglu A, Guven S, Imamoglu M. Contribution of MRI to ultrasound in the diagnosis of fetal anomalies. J Magn Reson Imaging. 2012 Apr;35(4):882-90. doi: 10.1002/jmri.23502. Epub 2011 Nov 29. PMID 22127893
- [Background] Prayer D, Brugger PC, Prayer L. Fetal MRI: techniques and protocols. Pediatr Radiol. 2004 Sep;34(9):685-93. doi: 10.1007/s00247-004-1246-0. Epub 2004 Jul 28. PMID 15316689
- [Background] Hill MC, Lande IM, Larsen JW Jr. Prenatal diagnosis of fetal anomalies using ultrasound and MRI. Radiol Clin North Am. 1988 Mar;26(2):287-307. PMID 3277224
- [Background] Jansz MS, Seed M, van Amerom JF, Wong D, Grosse-Wortmann L, Yoo SJ, Macgowan CK. Metric optimized gating for fetal cardiac MRI. Magn Reson Med. 2010 Nov;64(5):1304-14. doi: 10.1002/mrm.22542. PMID 20632406
- [Background] Saleem SN. Feasibility of MRI of the fetal heart with balanced steady-state free precession sequence along fetal body and cardiac planes. AJR Am J Roentgenol. 2008 Oct;191(4):1208-15. doi: 10.2214/AJR.07.3839. PMID 18806167
- [Background] Wedegartner U, Kooijman H, Yamamura J, Frisch M, Weber C, Buchert R, Huff A, Hecher K, Adam G. In vivo MRI measurement of fetal blood oxygen saturation in cardiac ventricles of fetal sheep: a feasibility study. Magn Reson Med. 2010 Jul;64(1):32-41. doi: 10.1002/mrm.22344. PMID 20572133
- [Background] Yamamura J, Kopp I, Frisch M, Fischer R, Valett K, Hecher K, Adam G, Wedegartner U. Cardiac MRI of the fetal heart using a novel triggering method: initial results in an animal model. J Magn Reson Imaging. 2012 May;35(5):1071-6. doi: 10.1002/jmri.23541. Epub 2012 Jan 13. PMID 22246623
- [Background] Lette J, Carini G, Tatum JL, Paquet N, Bisson G, Picard M, Bom HS, Lusa AM, Labanti G, Teitelbaum J, et al. Safety of dipyridamole testing in patients with cerebrovascular disease. Am J Cardiol. 1995 Mar 1;75(7):535-7. doi: 10.1016/s0002-9149(99)80602-x. No abstract available. PMID 7864009
- [Background] Nagel E, Lehmkuhl HB, Bocksch W, Klein C, Vogel U, Frantz E, Ellmer A, Dreysse S, Fleck E. Noninvasive diagnosis of ischemia-induced wall motion abnormalities with the use of high-dose dobutamine stress MRI: comparison with dobutamine stress echocardiography. Circulation. 1999 Feb 16;99(6):763-70. doi: 10.1161/01.cir.99.6.763. PMID 9989961
- [Background] Pennell DJ, Underwood SR, Ell PJ. Safety of dobutamine stress for thallium-201 myocardial perfusion tomography in patients with asthma. Am J Cardiol. 1993 Jun 1;71(15):1346-50. doi: 10.1016/0002-9149(93)90553-o. PMID 8498379
- [Background] Pennell DJ, Underwood SR, Manzara CC, Swanton RH, Walker JM, Ell PJ, Longmore DB. Magnetic resonance imaging during dobutamine stress in coronary artery disease. Am J Cardiol. 1992 Jul 1;70(1):34-40. doi: 10.1016/0002-9149(92)91386-i. PMID 1615867
- [Background] van Rugge FP, van der Wall EE, de Roos A, Bruschke AV. Dobutamine stress magnetic resonance imaging for detection of coronary artery disease. J Am Coll Cardiol. 1993 Aug;22(2):431-9. doi: 10.1016/0735-1097(93)90047-5. PMID 8335812
- [Background] Strigl S, Beroukhim R, Valente AM, Annese D, Harrington JS, Geva T, Powell AJ. Feasibility of dobutamine stress cardiovascular magnetic resonance imaging in children. J Magn Reson Imaging. 2009 Feb;29(2):313-9. doi: 10.1002/jmri.21639. PMID 19161182
- [Background] Hundley WG, Hamilton CA, Thomas MS, Herrington DM, Salido TB, Kitzman DW, Little WC, Link KM. Utility of fast cine magnetic resonance imaging and display for the detection of myocardial ischemia in patients not well suited for second harmonic stress echocardiography. Circulation. 1999 Oct 19;100(16):1697-702. doi: 10.1161/01.cir.100.16.1697. PMID 10525488
- [Background] Secknus MA, Marwick TH. Evolution of dobutamine echocardiography protocols and indications: safety and side effects in 3,011 studies over 5 years. J Am Coll Cardiol. 1997 May;29(6):1234-40. doi: 10.1016/s0735-1097(97)00039-9. PMID 9137218
- [Background] Hand JW, Li Y, Thomas EL, Rutherford MA, Hajnal JV. Prediction of specific absorption rate in mother and fetus associated with MRI examinations during pregnancy. Magn Reson Med. 2006 Apr;55(4):883-93. doi: 10.1002/mrm.20824. PMID 16508913
- [Background] Hand JW, Li Y, Hajnal JV. Numerical study of RF exposure and the resulting temperature rise in the foetus during a magnetic resonance procedure. Phys Med Biol. 2010 Feb 21;55(4):913-30. doi: 10.1088/0031-9155/55/4/001. Epub 2010 Jan 20. PMID 20090188
- [Background] De Wilde JP, Rivers AW, Price DL. A review of the current use of magnetic resonance imaging in pregnancy and safety implications for the fetus. Prog Biophys Mol Biol. 2005 Feb-Apr;87(2-3):335-53. doi: 10.1016/j.pbiomolbio.2004.08.010. PMID 15556670
- [Background] Chen MM, Coakley FV, Kaimal A, Laros RK Jr. Guidelines for computed tomography and magnetic resonance imaging use during pregnancy and lactation. Obstet Gynecol. 2008 Aug;112(2 Pt 1):333-40. doi: 10.1097/AOG.0b013e318180a505. PMID 18669732
- [Background] Shaikh MS, Lombay B. Fetal MRI : reviewing the history, indications, technique, safety and drawbacks. J Coll Physicians Surg Pak. 2004 Sep;14(9):576-9. PMID 15353148
- [Background] Haustein J, Laniado M, Niendorf HP, Louton T, Beck W, Planitzer J, Schoffel M, Reiser M, Kaiser W, Schorner W, et al. Triple-dose versus standard-dose gadopentetate dimeglumine: a randomized study in 199 patients. Radiology. 1993 Mar;186(3):855-60. doi: 10.1148/radiology.186.3.8430199.
- [Background] Niendorf HP, Alhassan A, Geens VR, Clauss W. Safety review of gadopentetate dimeglumine. Extended clinical experience after more than five million applications. Invest Radiol. 1994 Jun;29 Suppl 2:S179-82. doi: 10.1097/00004424-199406001-00059. No abstract available. PMID 7928222
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423
- [Background] Niendorf HP, Haustein J, Cornelius I, Alhassan A, Clauss W. Safety of gadolinium-DTPA: extended clinical experience. Magn Reson Med. 1991 Dec;22(2):222-8; discussion 229-32. doi: 10.1002/mrm.1910220212. PMID 1812350
- [Background] Niendorf HP, Haustein J, Louton T, Beck W, Laniado M. Safety and tolerance after intravenous administration of 0.3 mmol/kg Gd-DTPA. Results of a randomized, controlled clinical trial. Invest Radiol. 1991 Nov;26 Suppl 1:S221-3; discussion S232-5. doi: 10.1097/00004424-199111001-00075. No abstract available. PMID 1808134
- [Background] Dillman JR, Ellis JH, Cohan RH, Strouse PJ, Jan SC. Frequency and severity of acute allergic-like reactions to gadolinium-containing i.v. contrast media in children and adults. AJR Am J Roentgenol. 2007 Dec;189(6):1533-8. doi: 10.2214/AJR.07.2554. PMID 18029897
- [Background] Sundgren PC, Leander P. Is administration of gadolinium-based contrast media to pregnant women and small children justified? J Magn Reson Imaging. 2011 Oct;34(4):750-7. doi: 10.1002/jmri.22413. PMID 21928308
- [Background] Deo A, Fogel M, Cowper SE. Nephrogenic systemic fibrosis: a population study examining the relationship of disease development to gadolinium exposure. Clin J Am Soc Nephrol. 2007 Mar;2(2):264-7. doi: 10.2215/CJN.03921106. Epub 2007 Feb 7. PMID 17699423
- [Background] Mertes H, Sawada SG, Ryan T, Segar DS, Kovacs R, Foltz J, Feigenbaum H. Symptoms, adverse effects, and complications associated with dobutamine stress echocardiography. Experience in 1118 patients. Circulation. 1993 Jul;88(1):15-9. doi: 10.1161/01.cir.88.1.15. PMID 8319327
- [Background] Cicatiello AM, Landino P, Simonelli P, Del Mastro L, Ferrara P, Cioppa A, Ciaburri F. Safety of echo-dipyridamole test in elderly patients with coronary artery disease. Angiology. 1995 Apr;46(4):321-6. doi: 10.1177/000331979504600406. PMID 7726452
- [Background] Zaman M, Hashmi R, Niaz K, Ahmad A, Kamal S. Safety of pharmacological (intravenous dipyridamole) stress for Thallium-201 perfusion imaging in patients with coronary artery disease unable to exercise. J Pak Med Assoc. 1994 Oct;44(10):237-9. PMID 7815687
- [Background] Hunt CH, Hartman RP, Hesley GK. Frequency and severity of adverse effects of iodinated and gadolinium contrast materials: retrospective review of 456,930 doses. AJR Am J Roentgenol. 2009 Oct;193(4):1124-7. doi: 10.2214/AJR.09.2520. PMID 19770337
- [Background] Jeste DV, Palmer BW, Appelbaum PS, Golshan S, Glorioso D, Dunn LB, Kim K, Meeks T, Kraemer HC. A new brief instrument for assessing decisional capacity for clinical research. Arch Gen Psychiatry. 2007 Aug;64(8):966-74. doi: 10.1001/archpsyc.64.8.966. PMID 17679641
- [Result] Sarikouch S, Koerperich H, Boethig D, Peters B, Lotz J, Gutberlet M, Beerbaum P, Kuehne T. Reference values for atrial size and function in children and young adults by cardiac MR: a study of the German competence network congenital heart defects. J Magn Reson Imaging. 2011 May;33(5):1028-39. doi: 10.1002/jmri.22521. PMID 21509858
- [Derived] Olivieri LJ, Jiang J, Hamann K, Loke YH, Campbell-Washburn A, Xue H, McCarter R, Cross R. Normal right and left ventricular volumes prospectively obtained from cardiovascular magnetic resonance in awake, healthy, 0- 12 year old children. J Cardiovasc Magn Reson. 2020 Feb 3;22(1):11. doi: 10.1186/s12968-020-0602-z. PMID 32013998